CLINICAL TRIAL: NCT04952545
Title: A Phase 1 Study to Determine the Safety, Tolerability, and Pharmacokinetics of ALXN2050 in Healthy Participants of Japanese Descent
Brief Title: Study of ALXN2050 in Healthy Adult Participants of Japanese Descent
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: ALXN2050-HV-113
Record Dates: First submitted 2021-06-28; First posted 2021-07-07 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Healthy
Keywords: ALXN2050; Pharmacokinetics; Pharmacodynamics; Japanese Descent
MeSH Terms: interventions — rhoA GTP-Binding Protein

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: ALXN2050 (Dose 1) (Experimental): Participants will receive ALXN2050 (Dose 1) as follows under fasting conditions: 120-milligrams (mg) single dose, 3-day washout, then 120-mg twice daily (BID) dosing.
  Interventions: Drug: ALXN2050
- Cohort 1: Placebo (Dose 1) (Experimental): Participants will receive placebo (Dose 1) as follows under fasting conditions: 120-mg placebo single dose, 3-day washout, then 120-mg placebo BID dosing.
  Interventions: Drug: Placebo
- Cohort 2: ALXN2050 (Dose 2) (Experimental): Participants will receive ALXN2050 (Dose 2) as follows under fasting conditions: 180-mg single dose, 3-day washout, then 180-mg BID dosing.
  Interventions: Drug: ALXN2050
- Cohort 2: Placebo (Dose 2) (Experimental): Participants will receive placebo (Dose 2) as follows under fasting conditions: 180-mg placebo single dose, 3-day washout, then 180-mg placebo BID dosing.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALXN2050 — Oral tablet.
  Other Names: ACH-0145228 (formerly)
  Arms: Cohort 1: ALXN2050 (Dose 1); Cohort 2: ALXN2050 (Dose 2)
Drug: Placebo — Oral tablet.
  Arms: Cohort 1: Placebo (Dose 1); Cohort 2: Placebo (Dose 2)

SUMMARY:
This is a Phase 1 bridging study being conducted to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of ALXN2050 after both single- and multiple-dosing in healthy participants of Japanese descent.

ELIGIBILITY:
Key Inclusion Criteria:

* Medically healthy with no clinically significant or relevant abnormalities as determined by medical history, physical or neurological examination, vital signs, 12-lead electrocardiogram, screening clinical laboratory profiles.
* Participants must be of Japanese descent defined as:

  * First generation (born to 2 Japanese parents and 4 Japanese grandparents);
  * Born in Japan, and not have lived outside Japan for greater than 5 years;
  * Lifestyle, including diet, must not have significantly changed since leaving Japan.
* Participants must be able to speak, read, and understand the Japanese and English languages.
* Body mass index within the range 18.5 to 30.0 kilograms (kg)/meter squared, inclusive, with a minimum body weight of 50.0 kg at Screening.

Key Exclusion Criteria:

* History of any medical or psychiatric condition or disease that, in the opinion of the Investigator or designee, might limit the participant's ability to complete or participate in this clinical study, confound the results of the study, or pose an additional risk to the participant by their participation in the study.
* History of significant multiple and/or severe allergies.
* Any previous procedure that could alter absorption or excretion of orally administered drugs.
* Participation in another investigational drug or investigational device study within 5 half-lives (if known) or 30 days prior to the first dose of study intervention, whichever is longer.
* Body temperature ≥ 38.0°Celcius, at Screening or prior to the first dose of study intervention.
* History of drug or alcohol abuse within 2 years prior to the first dose of study intervention or positive drugs-of-abuse or alcohol screen at Screening or Day -1; current tobacco/nicotine users or smokers or a positive cotinine test at Screening.
* Donation of whole blood from 3 months prior to the first dose of study intervention, or of plasma from 30 days prior to the first dose of study intervention; receipt of blood products within 6 months prior to the first dose of study intervention.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-07-09 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2021-09-07 (Actual)

PRIMARY OUTCOMES:
Number Of Participants With Treatment-emergent Adverse Events | Day 1 (after first dose) through follow-up (7 +/- 2 days after final dose)
  see Time Frame - defined
Area Under The Concentration-time Curve From Time Zero To Infinity (AUCinf) For Single-dose ALXN2050 | Up to 72 hours postdose
  see Time Frame - defined
Maximum Plasma Concentration (Cmax) For Single-dose ALXN2050 | Up to 72 hours postdose
  see Time Frame - defined
Time To Maximum Plasma Concentration (Tmax) For Single-dose ALXN2050 | Up to 72 hours postdose
  see Time Frame - defined
Area Under The Concentration-time Curve From Time Zero To The 12-hour Time Point (AUC0-12) For Multiple-dose ALXN2050 | Up to 72 hours postdose
  see Time Frame - defined
Cmax For Multiple-dose ALXN2050 | Up to 72 hours postdose
  see Time Frame - defined
Tmax For Multiple-dose ALXN2050 | Up to 72 hours postdose
  see Time Frame - defined

SECONDARY OUTCOMES:
Alternative Pathway Activity As Measured By Wieslab Assay | Up to 72 hours postdose
  see Time Frame - defined
Complement Factor B Fraction b Levels | Up to 72 hours postdose
  see Time Frame - defined

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Site, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No